CLINICAL TRIAL: NCT06819631
Title: Retrospective and Observational Study in Relation to the Subjective Pain of Patients Attending the Corneal and Ocularcsurface Analysis Laboratory (LACSO) Affected by Ocular Surface Dysfunctions
Brief Title: Characterization of Subjective Discomfort in Patients With Tear Dysfunction
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: OFTAFONTANA_LACSO
Record Dates: First submitted 2025-01-10; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-10

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Characterization of subjective discomfort/pain in patients with ocular surface dysfunction in association with clinical and laboratory parameters, for a better understanding of the underlying pathogenic mechanisms.

DETAILED DESCRIPTION:
Dry Eye Disease (DED) is a multifactorial chronic disease impairing the ocular surface.

DED can be associated with conditions of inflammation and neurosensory dysfunction.

The aim of this study is to characterize the discomfort/pain in subjects affected by DED with the administration of scales, questionnaires, and analysis of corneal sensitivity by keratoesthesiometry, in association with clinical laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with suspected or diagnosed DED

Exclusion Criteria:

* nothing

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants in the study are patients suffering from ocular disconfort who are referred by their doctors for second/third level diagnostic tests at the University Ophthalmology Department. Patients are adults of both sexes, with eventual concomitant systemic and other ocular pathologies, without any limitation that defines exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Discomfort in subjects affected by Dry Eye Disease (DED) | Baseline (enrollment visit)
  Assessment of discomfort with Ocular Surface Disease Index (OSDI) and Dry Eye Questionaire-5 (DEQ-5)
Pain in subjects affected by Dry Eye Disease (DED) | Baseline (enrollment visit)
  Assessment of pain with Visual Analogue Scale (VAS) and Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Fontana, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy